CLINICAL TRIAL: NCT02219607
Title: Liver Enzymes and Fluid Balance Following Colorectal Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Pandazi Ageliki, Assistant Professor, Attikon Hospital
Other Study IDs: colorectal 1
Record Dates: First submitted 2014-08-16; First posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-08

CONDITIONS: Fluid Balance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- epidural
- general anesthesia

SUMMARY:
The use of epidural anesthesia and postoperative analgesia influences fluid balance following colorectal surgery.

Markers such as BNP (brain natriuretic peptide) and liver function enzymes can estimate intravascular fluid load and predict outcome after colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing colorectal surgery

Exclusion Criteria:

* Severe cardiac failure Severe renal failure Severe liver failure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients undergoing colorectal surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Change in liver enzymes | 5 days postoperatively

SECONDARY OUTCOMES:
Change in BNP (brain natriuretic peptide) | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Attikon Hospital, Chaïdári, Greece